CLINICAL TRIAL: NCT01678573
Title: A Single-Dose, Randomized, Open-Label, Three-Way Crossover Study to Evaluate the Pharmacokinetics of Abiraterone in Chinese Healthy Male Subjects
Brief Title: A Study to Evaluate the Pharmacokinetics of Abiraterone in Healthy Chinese Male Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR100668; ABI-PRO-1016 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2012-08-31; First posted 2012-09-05 (Estimated); Last update posted 2013-09-06 (Estimated); Status verified 2013-09

CONDITIONS: Healthy
Keywords: Healthy; Pharmacokinetics; Abiraterone acetate; Abiraterone; JNJ-212082; Zytiga; Chinese; Fasted
MeSH Terms: interventions — Abiraterone Acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sequence 1: abiraterone acetate (Experimental): Randomly assigned participants in Sequence 1 will receive different dose levels of abiraterone acetate (Treatment A = 250 mg; Treatment B = 500 mg; and Treatment C = 1000 mg) on Day 1 in each of the 3 treatment periods according to the randomized schedule "ABC" under fasted conditions.
  Interventions: Drug: Treatment A: abiraterone acetate; Drug: Treatment B: abiraterone acetate; Drug: Treatment C: abiraterone acetate
- Sequence 2: abiraterone acetate (Experimental): Randomly assigned participants in Sequence 2 will receive different dose levels of abiraterone acetate (Treatment A = 250 mg; Treatment B = 500 mg; and Treatment C = 1000 mg) on Day 1 in each of the 3 treatment periods according to the randomized schedule "BAC" under fasted conditions.
  Interventions: Drug: Treatment A: abiraterone acetate; Drug: Treatment B: abiraterone acetate; Drug: Treatment C: abiraterone acetate
- Sequence 3: abiraterone acetate (Experimental): Randomly assigned participants in Sequence 3 will receive different dose levels of abiraterone acetate (Treatment A = 250 mg; Treatment B = 500 mg; and Treatment C = 1000 mg) on Day 1 in each of the 3 treatment periods according to the randomized schedule "CBA" under fasted conditions.
  Interventions: Drug: Treatment A: abiraterone acetate; Drug: Treatment B: abiraterone acetate; Drug: Treatment C: abiraterone acetate

INTERVENTIONS:
Drug: Treatment A: abiraterone acetate — 250 mg/day tablet administered orally on Day 1 of each treatment period.
  Other Names: ZYTIGA
Drug: Treatment B: abiraterone acetate — 500 mg/day tablets administered orally on Day 1 of each treatment period.
  Other Names: ZYTIGA
Drug: Treatment C: abiraterone acetate — 1000 mg/day tablets administered orally on Day 1 of each treatment period.
  Other Names: ZYTIGA

SUMMARY:
The purpose of this study is to evaluate the pharmacokinetics (how the drug concentrations change over time) of abiraterone acetate after oral administration of abiraterone acetate at different dose levels of 250, 500, and 1000 mg in healthy Chinese male participants under fasted conditions.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), randomized (the treatment sequence is assigned by chance), 3-way crossover study (method used to switch participants from one dose level to another in a clinical study) of single doses of abiraterone acetate in healthy Chinese male participants. The study consists of 3 phases: screening, open-label treatment, and follow up phases. After screening, randomly assigned participants will receive different dose levels of abiraterone acetate (Treatment A = 250 mg; Treatment B = 500 mg; and Treatment C = 1000 mg) on Day 1 in each of the 3 treatment periods according to a randomized schedule under fasted conditions (Sequence 1 = ABC; Sequence 2 = BAC; and Sequence 3 = CBA). Each treatment period will be separated by a washout period (period when participant is not receiving any study medication) of at least 7 days. In the follow-up phase, study-related adverse events will be monitored by the investigator. Serial blood samples for pharmacokinetic analysis will be collected and safety will be monitored throughout the study. The total study duration will be approximately 42 days.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index within 18 to 27 kg/m2 (inclusive) and body weight above 50 kg at screening
* Protocol-defined laboratory and electrocardiogram parameters
* Negative test results for selected medications and substances of abuse and negative exhaled carbon monoxide test at check-in day of each period
* Agrees to protocol-defined use of effective contraception
* Willing to be confined at the clinical research facility for time period specified in the protocol

Exclusion Criteria:

* Significant history or current manifestation of any significant metabolic, allergic, dermatological, hepatic, renal, hematologic, pulmonary, cardiovascular, gastrointestinal, neurological, or psychiatric disorder
* History of hypersensitivity reaction to the study medication or related compounds or excipients used in the formulation
* Confirmed hepatitis A, B, or C infection or human immunodeficiency virus (HIV) 1 or HIV-2 infection at screening
* Serum testosterone level of <200 ng/dL
* Use of any tobacco or nicotine-containing products
* Known or suspected use of illicit drugs in the last year
* Protocol contraindicated medications/preparations (prescription and non-prescription)

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2012-07; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Maximum observed plasma concentration of abiraterone | Pre-dose and up to 96 hours post-dose each treatment period
Time to reach the maximum observed plasma concentration of abiraterone | Pre-dose and up to 96 hours post-dose each treatment period
Area under the plasma concentration-time curve from time 0 to the last quantifiable concentration of abiraterone | Pre-dose and up to 96 hours post-dose each treatment period
Area under the plasma concentration-time curve extrapolated to infinite time of abiraterone | Pre-dose and up to 96 hours post-dose each treatment period
Apparent terminal elimination rate constant of abiraterone | Pre-dose and up to 96 hours post-dose each treatment period
Apparent terminal elimination half-life of abiraterone | Pre-dose and up to 96 hours post-dose each treatment period

SECONDARY OUTCOMES:
Number of participants with adverse events | Up to 42 days

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Beijing, China